CLINICAL TRIAL: NCT02862145
Title: A Multicenter Phase 1B Pharmacodynamics Study of MRX34, MicroRNA miR-Rx34 Liposomal Injection, in Patients With Advanced Melanoma and Biopsy Accessible Lesions
Brief Title: Pharmacodynamics Study of MRX34, MicroRNA Liposomal Injection in Melanoma Patients With Biopsy Accessible Lesions
Acronym: MRX34-102
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: 5 immune related serious adverse events in Phase 1 study
Sponsor: Mirna Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRX34-102
Record Dates: First submitted 2016-07-29; First posted 2016-08-10 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-07

CONDITIONS: Melanoma
Keywords: Biosy accessible melanoma
MeSH Terms: conditions — Melanoma | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with MRX34 (Experimental): Liposomal Injection of MRX34 for 5 days followed by 16 days rest with premedication of dexamethasone daily.
  Interventions: Drug: MRX34; Drug: Dexamethasone

INTERVENTIONS:
Drug: MRX34 — Treatment of melanoma with pharmacodynamics biopsy of tissue and blood
  Other Names: miR-Rx34
Drug: Dexamethasone — Premedication during the week of treatment
  Other Names: Decadron

SUMMARY:
This study is designed to investigate the biomarkers, pharmacodynamics and pharmacokinetics of the liposomal micro-ribonucleic acid-34 (microRNA-34, miR-34). Melanoma patients with easily accessible lesions will undergo serial biopsies and serial blood samples will be collected.

DETAILED DESCRIPTION:
MRX34 Induction Therapy consists of 3 cycles of MRX34 treatment given over an approximately 8 week period. Dexamethasone 10 mg PO (or IV) will be given as premedication. On Days 1-5 of each treatment cycle, MRX34 will be given as a daily infusion followed by 16 days of rest. At screening a tumor biopsy sample will be required from all patients. Additional biopsies will be collected at Cycle 1 Day 3 and the end of Cycles 1 and 3 (Day 18 +/- 1 day)

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Advanced or metastatic cutaneous, acral or mucosal melanoma
* Tumor lesions accessible to serial biopsies
* ECOG ≤ 1
* ANC ≥, Plts ≥100,000 /mm3

Exclusion Criteria:

* Serious active non-malignant disease
* Central Nervous System metastasis

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Peak blood concentration and Area Under the Curve (AUC) of MRX34 after IV dosing and drug concentration in tissue biopsies | 3 months

SECONDARY OUTCOMES:
Frequency and severity of adverse events associated with MRX34 treatment | 6 months

OTHER OUTCOMES:
Change in tumor measurements over time using RECIST criteria. | 6 months
RNA sequencing analysis of PBMCs to evaluate gene expression through TLR signaling, RIG-I Pathway and PD1/PD-L1 Blockade. | During 3 months of treatment
Assessment of MRX34 accumulation in tumor tissue measured by qPCR and CISH. | During 3 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Susan Smith, MSN, Study Director — Mirna Therapeutics

IPD SHARING:
Plan to Share IPD: No